CLINICAL TRIAL: NCT02398799
Title: Supporting Dyads Affected by Heart Failure - A Randomised Controlled Study Evaluating a Psychoeducational Intervention
Brief Title: Supporting Dyads Affected by Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anna Stroemberg, professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 03-568
Record Dates: First submitted 2015-03-08; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): The dyads in the control group received care as usual including traditional care in hospital and outpatient education and support. The care is mainly focused on the patient's needs. The partner is not systematically involved in the follow-up focusing on education and psychosocial support.
- Psycho edcuactional support (Experimental): The intervention psychoeducational support to the patient-partner dyads was delivered in 3 sessions through nurse-led face-to-face counseling, a computer-based CD-ROM program and other written teaching materials. All sessions lasted at least 60 minutes and were conducted in the dyads' homes or in the heart failure clinic. The first session 2 weeks after discharge and the two remaining sessions 6- and 12-weeks following discharge. Each session included education on heart failure and development of problem- solving skills to assist the dyads in recognizing and modifying factors that contribute to psychological and emotional distress. The intervention focused on changing thoughts and behaviors and implementing strategies for self-care.
  Interventions: Behavioral: Psychoeducational support

INTERVENTIONS:
Behavioral: Psychoeducational support — The intervention was based on a conceptual model from Stuifbergen. The model has sprung from Pender's model of health promotion and Bandura's self-efficacy theory. Cognitive-behavioral strategies were chosen to assist dyads in recognizing and modifying factors that contribute to physical and emotional distress by changing thoughts and behaviors and assisting dyads in solving problems related to implementing strategies for self-care.
  Shared care is a dyadic process based on the assumption that each participant affects and is affected by the other. Shared goals and a shared commitment provide the essential building blocks of the dyad relationship. The dyad structure presents an opportunity for healthcare professionals to integrate a collaborative patient-partner centered effort.
  Arms: Psycho edcuactional support

SUMMARY:
The aim of this randomized controlled trial was to evaluate the effects of an integrated dyad care program with education and psychosocial support to patients with chronic heart failure and their partners during a post-discharge period after acute deterioration of heart failure.

Methods: One hundred fifty five patient-caregiver dyads has been randomized to usual care or a psycho-education intervention delivered in three modules through nurse-led face-to-face counseling, computer-based education and other written teaching materials to assist dyads develop problem-solving skills. Follow-up assessments has been completed after 3, 12 and 24 months to assess perceived control, perceived health, depressive symptoms, self-care, knowledge, caregiver burden and health care utilization.

DETAILED DESCRIPTION:
Heart failure is a serious condition with a poor prognosis. It is the leading cause of hospitalization and readmissions for worsening heart failure remains high. Treatment aims to reduce symptoms and morbidity and to improve quality of life and survival. Counseling and education is an important part of treatment, but despite the fact that most patients receive education, many are not able to adequately engage in self-care activities. Non-adherence to self-care recommendations is high which may be a contributing factor for worsening heart failure and to the high number of readmissions.

Having support of a partner is important for patients with heart failure. Supportive others have the potential to improve self-care outcomes and increase adherence to treatment. At the same time, it should be acknowledged that the disease can also affect the partners negatively. However, emotional reactions of burden and stress decrease when partner's experiences control over the heart disease.

Despite the fact that heart failure has a number of negative consequences for patients and the partners, research addressing self-care barriers from a family perspective is rare, and until now contemporary care has remained patient focused. Previous studies have indicated the importance of partner support but have not found the appropriate methods for involving and encourage partners. Therefore, studies focusing on the heart failure patient-partner dyad are needed, but to date, most studies have only evaluated short term effects of intervention programs, while long term effects might be of equally importance. The aim of this randomized controlled study was to evaluate the effects of an integrated dyad care program with education and psychosocial support to patients with chronic heart failure and their partners during a post-discharge period after acute deterioration of heart failure.

Methods: One hundred fifty five patient-caregiver dyads has been randomized to usual care (n = 71) or a psycho-education intervention (n = 84) delivered in three modules through nurse-led face-to-face counseling, computer-based education and other written teaching materials to assist dyads develop problem-solving skills. Follow-up assessments has been completed after 3, 12 and 24 months to assess perceived control, perceived health, depressive symptoms, self-care, knowledge, caregiver burden and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were to be a dyad consisting of a patient diagnosed with heart failure based on the European Society of Cardiology guidelines,
* New York Heart Association (NYHA) class II-IV,
* with a partner living in the same household as the patient,
* recently discharged from hospital (i.e. 2-3 weeks) following a heart failure acute exacerbation.

Exclusion Criteria:

* Exclusion criteria for the dyads were dementia, or other severe psychiatric illnesses,
* drug abuse,
* difficulties in understanding or reading the Swedish language,
* undergoing cardiac surgery including cardiac transplant or
* participating in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-01; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Perceived control measure by Control Attitude Scale | 3 months
  Perceived control in patients and partners

SECONDARY OUTCOMES:
Quality of life measure by SF-36 | 3, 12 and 24 months
  Quality of life in patients and partners
Self care measured by European Self-care Behaviour Scale | 3, 12 and 24 months
  Self care in patients
Caregiverburden measured by Caregiverburden Scale | 3, 12 and 24 months
  Caregiverburden in partners

REFERENCES:
- [Derived] Liljeroos M, Agren S, Jaarsma T, Stromberg A. Dialogues between nurses, patients with heart failure and their partners during a dyadic psychoeducational intervention: a qualitative study. BMJ Open. 2017 Dec 14;7(12):e018236. doi: 10.1136/bmjopen-2017-018236. PMID 29247098
- [Derived] Liljeroos M, Agren S, Jaarsma T, Arestedt K, Stromberg A. Long-term effects of a dyadic psycho-educational intervention on caregiver burden and morbidity in partners of patients with heart failure: a randomized controlled trial. Qual Life Res. 2017 Feb;26(2):367-379. doi: 10.1007/s11136-016-1400-9. Epub 2016 Sep 8. PMID 27631892
- [Derived] Liljeroos M, Agren S, Jaarsma T, Arestedt K, Stromberg A. Long Term Follow-Up after a Randomized Integrated Educational and Psychosocial Intervention in Patient-Partner Dyads Affected by Heart Failure. PLoS One. 2015 Sep 25;10(9):e0138058. doi: 10.1371/journal.pone.0138058. eCollection 2015. PMID 26406475